CLINICAL TRIAL: NCT06683872
Title: Evaluation of Clinical Efficacy and Prognosis in Patients with Hypertrophic Obstructive Cardiomyopathy Through Hemodynamic Modeling Reconstructed by CT
Status: Enrolling by invitation | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024113
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: Hypertrophic cardiomyopathy; computational fluid dynamics
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with hypertrophic cardiomyopathy undergoing septal reduction therapy.
  Interventions: Procedure: surgical myectomy

INTERVENTIONS:
Procedure: surgical myectomy — Our procedure was performed via a right infra-axillary incision (4-5 cm), enter the thoracic cavity through the third intercostal space lateral to the pectoralis major muscle. Generally, neither rib resection nor division of the pectoralis major muscle were required. The intervention utilized femoral-femoral cardiopulmonary bypass (CPB). The aorta was clamped using a Glauber clamp (CardioVision MICAortic Clamp, Cardiomedical GmbH). Myocardial protection was achieved with antegrade Del Nido cardioplegia. After inducing of cardiac asystole, a transverse incision was made in the aorta and the aorta incision was suspended to enhance visualization. A mesh retractor (FEHLING INSTRUMENTS, Karlstein, Germany) was placed in the aortic sinus to protect the aortic leaflets. The extent of the septal myectomy, determined based on preoperative TEE, started 5 mm below the midpoint of the right coronary cusp. It extended counterclockwise towards the anterior commissure of the mitral valve a

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a common autosomal dominant inherited heart disease, with previous data suggesting a prevalence of approximately 1 in 500 in the population. However, with the widespread use of genetic testing and high-sensitivity cardiac imaging in recent years, the estimated prevalence of HCM may be as high as 1 in 200. Approximately 75% of HCM patients will develop left ventricular outflow tract obstruction (LVOTO), leading to decreased exercise capacity, dyspnea, syncope, heart failure, and even sudden death, significantly impacting the patients' quality of life and survival.

The optimal treatment for hypertrophic obstructive cardiomyopathy (HOCM) is still a matter of controversy, despite surgical myectomy being considered the "gold standard" for HOCM treatment. Treatment options such as chemical (radiofrequency) ablation and medications (Mavacamten) are also challenging the status, and there is even debate over the surgical approach for myectomy. Currently, there is no consensus in the medical community about the pathophysiological mechanisms of LVOTO, and the exact mechanisms of its occurrence are not fully understood, which is also a major reason for the treatment controversy in HOCM patients.

The focus of clinical decision-making is on the treatment based on the LVOTO pressure gradient, and it is generally recommended internationally to consider invasive treatment when the LVOTO pressure gradient is ≥50mmHg. However, there are still a small number of patients who do not have symptoms with a pressure gradient greater than 50mmHg or have significant symptoms with a pressure gradient less than 50mmHg, indicating that relying solely on the pressure gradient to assess the severity of HOCM and its prognosis may not be comprehensive enough.

In recent years, with the development of medical engineering integration, the use of computational fluid dynamics (CFD) in the medical field, particularly in the field of cardiovascular diseases, has become increasingly widespread. CFD can construct cardiovascular geometric models based on specific clinical images of a patient and simulate ventricular wall motion and blood flow within the heart through computer calculations to obtain the required hemodynamic parameters. This enables the visualization and quantification of intraventricular blood flow. Compared to direct measurement techniques based on imaging, CFD has advantages such as non-invasiveness, comprehensiveness, and accuracy, leading to its increasing application in cardiovascular function research. In particular, in the field of cardiomyopathy, CFD can help deepen the understanding of the pathophysiological mechanisms of hypertrophic obstructive cardiomyopathy by reconstructing the anatomical configuration of the left ventricle and analyzing intraventricular blood flow and related hemodynamic parameters, which in turn can aid in clinical decision-making and the assessment of clinical prognosis. Therefore, we propose using three-dimensional (3D) computed tomography (CT) simulation technology to assess the hemodynamics of patients with hypertrophic obstructive cardiomyopathy, in order to guide clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-70 years old 2. Maximum interventricular septum thickness ≥15mm 3. Dynamic left ventricular outflow tract gradient at rest or with provocation (Valsalva maneuver or exercise) ≥50mmHg 4. New York Heart Association (NYHA) functional classification ≥II 5. Presence of severe symptoms despite maximal medical therapy (maximal medical therapy for HCM may include combination of disopyramide and/or β-blockers and calcium channel blockers)

Exclusion Criteria:

* 1. Combined with other heart diseases that require surgical treatment, such as heart valve disease or coronary artery atherosclerotic heart disease.

  2. Left ventricular ejection fraction <40%. 3. Presence of the following arrhythmias: atrial fibrillation, QT interval > 500ms, occurrence of sustained ventricular tachycardia in the past 6 months before screening.

  4. Allergy to iodine contrast agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient diagnosed with hypertrophic cardiomyopathy comes from the Zhejiang Province People's Hospital, the First Affiliated Hospital of Shanghai Jiaotong University School of Medicine, and the Second Affiliated Hospital of Nanchang University.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in left ventricular outflow tract pressure immediately after surgery and at 1 year postoperatively | From operation to one year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Province People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Houston BA, Stevens GR. Hypertrophic cardiomyopathy: a review. Clin Med Insights Cardiol. 2015 Jan 26;8(Suppl 1):53-65. doi: 10.4137/CMC.S15717. eCollection 2014. PMID 25657602